CLINICAL TRIAL: NCT06632483
Title: Retrospective, Non-interventional Database Study for the Evaluation of Real-world Drug Use Patterns, Clinical Characteristics and Clinical Outcomes in Patients Initiated on Vericiguat in India
Brief Title: An Observational Study to Learn More About How Safe Vericiguat is and How Well it Works in Indian People With Chronic Heart Failure With Reduced Ejection Fraction and Worsening Chronic Heart Failure Under Real World Conditions
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22613
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction; Worsening Chronic Heart Failure
Keywords: HFrEF
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vericiguat: New users who have been initiated on Vericiguat between 01 Sep 2022 and 31 Aug 2023 in 15 Sites in India
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Prescibed as per local label

SUMMARY:
This is an observational study in which data already collected from people with chronic HFrEF (heart failure with reduced ejection fraction) who have experienced worsening heart failure are studied.

Chronic HFrEF is a long-term condition where the left side of the heart does not pump blood out to the body as well as it should. Blood and fluid may collect in the lungs, blood vessels, and tissues causing shortness of breath or tiredness. Over time, heart failure can lead to other serious medical conditions that may result in hospital stays and even death.

The study drug, vericiguat, is already approved for doctors to prescribe to people with worsening of heart failure with chronic HFrEF in India.

Vericiguat increases the activity of an enzyme called soluble guanylate cyclase (sGC), which relaxes the blood vessels, allowing more blood to flow through. As a result, the heart is able to pump better.

The participants in this study are already receiving treatment with vericiguat as part of their regular care from their doctors. There is currently limited real-world data on the use of vericiguat. Furthermore, discussing whether vericiguat treatment should start early in people with heart failure can help doctors manage these people better.

The main purpose of this study is to collect information about how well vericiguat works and how safe it is in Indian people with chronic HFrEF who have experienced worsening heart failure. To do this, researchers will collect the following information:

* participants' characteristics, including age, sex, height, weight, and medical history
* additional medicines participants have taken with vericiguat
* other treatment options participants have taken for the treatment of heart failure
* levels of NT-pro BNP* in participants' blood at least one month before taking vericiguat (*NT-proBNP is made by heart muscles. People with heart diseases have increased levels of NT-proBNP in their blood. Measuring NT-proBNP levels in the blood can help doctors identify heart disease.)
* number of participants from India, divided into four zones-North, South, East, and West
* categorization of participants based on how heart failure limits physical activity and classification of heart failure by cause
* change in heart function measured by how much blood the left side of the heart can pump out
* number of hospitalizations and number of participants who died due to heart-related and non-heart-related events
* number of participants who experienced low blood pressure or fainting after starting treatment with vericiguat
* participants who discontinued treatment with vericiguat, due to low blood pressure or fainting

The data will come from the participants' hospital, medical and electronic healthcare records. Data collected will be from Indian people with chronic HFrEF who started taking vericiguat between September 2022 and August 2023.

Researchers will track participants' data and will follow them until Feb 2024. In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ≥18 years age.
* Patients who are prescribed as per local label will be included in the study
* At least one Vericiguat prescription during the time between 01 Sep 2022 and 31 Aug 2023

Exclusion Criteria:

* Subjects who have participated in an interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary source of data is hospital medical records. The electronic health records or physical records of patients with HFrEF who were managed with Vericiguat will be screened to obtain the relevant baseline and follow-up data. Such records will be collected from 15 participating sites in India.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive measurement of baseline clinical characteristics of patients initiated on Vericiguat | At baseline
  Clinical characteristics include demographics, concomitant medication, medical history and surgical history, history of hospitalization, N-Terminal Pro Brain Natriuretic Peptide (NT-Pro BNP) levels
Descriptive measurement of baseline treatment patterns of patients initiated on Vericiguat | At baseline
Description of the use of medications of interest (yes/no) before/after initiation of Vericiguat | Up to 12 months
  Includes description of prescribed amount of medications of interest in respective observation periods
Descriptive measurement of titration patterns | Up to 12 months
  Includes starting dose, up-titration / down-titration (yes/no), time until target dose
Descriptive measurement of treatment discontinuation | Up to 12 months
  Includes descriptive analysis of number of patients who have discontinued treatment, time points of discontinuation, reasons for discontinuation (Symptomatic hypotension, syncope)

SECONDARY OUTCOMES:
Number of patients with hospitalizations due to heart failure after Vericiguat initiation | Up to 12 months
Cardiovascular mortality rate | Up to 12 months
Composite of heart failure hospitalization and cardiovascular mortality | Up to 12 months
Number of patients with symptomatic hypotension or syncope after Vericiguat initiation | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.